CLINICAL TRIAL: NCT04006145
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Study to Explore the Efficacy and Safety of Elobixibat in Adults With Nonalcoholic Fatty Liver Disease (NAFLD) or Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Phase 2 Study of Elobixibat in Adults With NAFLD or NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3309-012
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — elobixibat

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Placebo-Controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elobixibat (Experimental): Elobixibat 5 mg once daily
  Interventions: Drug: Elobixibat
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Elobixibat — Elobixibat is a small molecule and a potent inhibitor of the ileal bile acid transporter (iBAT).
  Other Names: A3309
  Arms: Elobixibat
Drug: Placebo oral tablet — Placebo identical in appearance to active drug
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Double-blind, randomized, placebo-controlled study to explore the efficacy and safety of elobixibat compared to placebo in adults with NAFLD (nonalcoholic fatty liver disease) or NASH (nonalcoholic steatohepatitis)

DETAILED DESCRIPTION:
A total of 15 investigators at 15 sites received institutional review board (IRB)/ethics committee (EC) approval to participate in this study and enrolled at least 1 participant.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a current biopsy-confirmed NASH within 6 months of screening or a suspected diagnosis of NAFLD/NASH
* Screening magnetic resonance imaging-proton density fat fraction (MRI-PDFF) with ≥10% liver steatosis
* Fasting serum low density lipoprotein-cholesterol (LDL-C) >130 mg/dL at Screening, >110 mg/dL on lipid-lowering medications

Key Exclusion Criteria:

* Body mass index (BMI) <25 kg/m2
* Fibrosis-4 index (Fib-4) >2.6
* Any of the following laboratory abnormalities:

  1. alanine aminotransferase (ALT) >5 × upper limit of normal (ULN) or aspartate aminotransferase (AST) >5 × ULN
  2. International normalized ratio (INR) ≥1.3, unless on anticoagulant therapy
  3. Total bilirubin >ULN, except with an established diagnosis of Gilbert's syndrome
  4. Platelet count less than the lower limit of normal (LLN)
  5. Creatinine clearance as calculated by the modification of diet in renal disease (MDRD) estimated glomerular filtration rate (eGFR) equation <60 mL/min
* Uncontrolled Type 2 diabetes defined as hemoglobin A1c (HbA1c) >9.5%
* Clinical hyperthyroidism or hypothyroidism or screening hormone results pointing to thyroid dysfunction.
* Uncontrolled hypertension
* Participants with known intolerance to MRI or with conditions contraindicated for MRI procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Hope Clinical Research, Canoga Park, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Integrity Clinical Research, LLC, Doral, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Guardian Angel Research Center, Inc., Tampa, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind, randomized, placebo-controlled, phase 2 study was conducted at 15 sites in the United States to explore the efficacy and safety of elobixibat (oral dose of 5 milligrams [mg]) once daily for 16 weeks in participants with nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH).
Pre-assignment Details: The study consisted of a 6-week screening period followed by a 16-week treatment period and a follow-up visit 2 weeks after the last dose of study drug.
Period: Overall Study
Arm/Group | Elobixibat | Placebo
Started | 23 | 24
Received Treatment | 23 | 24
Completed | 22 | 21
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elobixibat | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.77) | 50.0 (13.36) | 50.9 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 3 | 0 | 3
  Race: Black or African American | 2 | 2 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 18 | 21 | 39
  Race: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47
Disease under study [Count of Participants; unit: Participants] — One participant was counted under both NAFLD and NASH per case report form (CRF) collected data.
  Participants
    Nonalcoholic Fatty Liver Disease (NAFLD) | 13 | 13 | 26
    Nonalcoholic Steatohepatitis (NASH) | 11 | 11 | 22
Duration of disease (Years) [Mean (Standard Deviation); unit: years] — Population: One participant was counted under both NAFLD and NASH per case report form (CRF) collected data.
  years
    Nonalcoholic Fatty Liver Disease (NAFLD): number analyzed (Participants) | 13 | 13 | 26
    Nonalcoholic Fatty Liver Disease (NAFLD) | 1.879 (2.667) | 1.534 (2.908) | 1.707 (2.739)
    Nonalcoholic Steatohepatitis (NASH): number analyzed (Participants) | 11 | 11 | 22
    Nonalcoholic Steatohepatitis (NASH) | 1.610 (2.918) | 0.892 (1.246) | 1.251 (2.220)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Low Density Lipoprotein-cholesterol (LDL-C) at Week 16
Description: The primary efficacy endpoint was the change from Baseline in serum LDL-C at Week 16. Baseline was defined as the last non-missing LDL-C value prior to the first dose of study drug.
Time Frame: Week 16
Population: The intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: "mmol/L"
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 23 | 24
"mmol/L" | -0.57 (0.125) | -0.17 (0.134)
Statistical Analysis 1: Comparison: Elobixibat vs Placebo; Change from baseline in serum LDL-C at Week 16 was analyzed using ANCOVA after the missing data imputation, with treatment group as a factor, baseline serum LDL-C, baseline LDL-C-by-treatment interaction values, and baseline lipid-lowering medications (Yes or No) as covariates. Missing data for serum LDL-C was imputed through multiple imputation method as described in the statistical analysis plan (SAP); Test type: Superiority; p = 0.029, ANCOVA; LS-Means Difference = -0.40, 95% CI 2-sided [-0.76 to -0.04], Standard Error of Mean 0.184

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in enrolled participant regardless of causal relationship with study drug. An SAE was defined as any AE that, at any dose, resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity, required or prolonged hospitalization, was a congenital anomaly/birth defect or an important medical event. TEAEs were defined as AEs that were new or worsened after the first dose of study drug.
Time Frame: From first dose of study drug (Day 1) up to end of follow-up per participant, approximately 13 months
Population: The safety population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 23 | 24
Participants
  TEAEs | 13 | 10
  TESAEs | 0 | 0

3. Secondary Outcome: Absolute Change From Baseline to Week 16 in Liver Fat Fraction
Description: The effect of elobixibat on liver steatosis was measured by magnetic resonance imaging (MRI) for liver fat fraction using proton density fat fraction [PDFF]). Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: The ITT population included all randomized participants who received at least 1 dose of study drug. Only those participants with data collected at Baseline and Week 16 are reported.
Measure: Least Squares Mean (Standard Error); unit: percent of liver fat
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 21 | 18
percent of liver fat | -0.43 (1.203) | 0.09 (1.299)

4. Secondary Outcome: Absolute Change From Baseline to Week 16 in Total Liver Fat
Description: The effect of elobixibat on liver steatosis was measured by MRI for total liver fat using whole liver fat volume. Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milliliter
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 21 | 18
milliliter | -2.80 (36.240) | 7.95 (39.146)

5. Secondary Outcome: Change From Baseline to Week 16 in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Gamma-glutamyl Transferase (GGT)
Description: Serum samples were collected at specified timepoints to assess ALT, AST and GGT levels. Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units/liter
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 22 | 20
Units/liter
  ALT | 5.04 (3.914) | 1.05 (3.969)
  AST | 2.21 (2.250) | 0.96 (2.359)
  GGT | 5.12 (2.009) | -1.73 (2.108)

6. Secondary Outcome: Change From Baseline to Week 16 in High-density Lipoprotein (HDL) Cholesterol, Non-high-density Lipoprotein Cholesterol and Triglycerides
Description: Blood samples were collected at specified timepoints to assess HDL and non-HDL cholesterol levels and triglycerides. Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 22 | 20
millimoles/liter
  HDL cholesterol | 0.03 (0.047) | -0.05 (0.049)
  Non-HDL cholesterol | -0.75 (0.154) | -0.23 (0.162)
  Triglycerides | -0.13 (0.149) | -0.08 (0.156)

7. Secondary Outcome: Change From Baseline to Week 16 in Low-density Lipoprotein (LDL) Cholesterol to High-density Lipoprotein Cholesterol Ratio
Description: Blood samples were collected at specified timepoints to assess LDL and HDL cholesterol levels and ratio was obtained. Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 22 | 20
ratio | -0.56 (0.158) | -0.11 (0.166)

8. Secondary Outcome: Change From Baseline to Week 16 in Total Bile Acids
Description: Blood samples were collected at specified timepoints to assess total bile acid levels. Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: micromoles/liter
Arm/Group | Elobixibat | Placebo
Number analyzed (Participants) | 22 | 20
micromoles/liter | 0.49 (0.696) | 0.33 (0.714)

ADVERSE EVENTS:
Time Frame: Adverse events and deaths were collected from first dose of study drug (Day 1) up to end of follow-up per participant, approximately 13 months
Description: Analysis was performed on the safety analysis set.
Arm/Group | Elobixibat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 13/23 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elobixibat (N=23) | Placebo (N=24)
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Bacterial abdominal infection (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Albireo will retain the ownership of all data. All proposed publications based on this study must be subject to the sponsor's approval requirements.

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04006145/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT04006145/SAP_001.pdf